CLINICAL TRIAL: NCT00426192
Title: Mechanisms of Endotoxin-Tolerance of Human Monocytes After CABG-Sugery - Effects of Hemofiltration and Mannitol Treatment
Brief Title: Effects of Hemofiltration and Mannitol Treatment on Cardiopulmonary-Bypass Induced Immunosuppression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Saarland (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AN-01
Record Dates: First submitted 2007-01-03; First posted 2007-01-24 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Inflammation
Keywords: Immunedefense Suppression; Cardiopulmonary Bypass; Mannitol; Hemofiltration; Cytokines; Receptors, Surface CD14
MeSH Terms: conditions — Inflammation | interventions — Hemofiltration

INTERVENTIONS:
Drug: i.v. mannitol
Procedure: hemofiltration

SUMMARY:
After cardiac surgery with cardiopulmonar bypass, the LPS-stimulated cytokine response has been previously shown to be depressed. Therefore, in this trial the hypothesis was tested, whether simple immunomodulting interventions like the i.v. adminstration of mannitol of hemofiltration during cardipulmonary bypass can attenuate this immunosuppressing effect.

DETAILED DESCRIPTION:
Background Cardiac surgery using cardiopulmonary bypass (CPB) causes a systemic inflammatory response. In addition to this immune response to CPB, a significant impairment of the responsiveness of peripheral blood mononuclear cells (PBMC) to further immunological stimuli has been observed. The aim of our present study was to evaluate the ability of antioxidant therapy with mannitol or hemofiltration during CPB to modulate the observed immunosuppression after CPB.

Methods With ethics committee approval, 52 patients undergoing elective CABG-surgery were prospectively enrolled and randomized into 3 groups (control, 50 g mannitol iv, hemofiltration during CPB). Blood samples were taken after induction of anesthesia (T1), 20 min after separation from CPB (T2) and 24 h postoperatively (T3). Expression density of the monocytic surface receptor CD14, HLA-DR expression and cytokine release (TNF- and IL10) after LPS-stimulation were evaluated.

Results At T2, the CD14dim cell population was maintained in both intervention groups while in the control group there was a significant decrease of this proinflammatory monocytic phenotype. At T3, all groups developed a significant shift towards the antiinflammatory CD14bright population. No significant differences regarding HLA-DR expression or cytokine release could be demonstrated.

Conclusion This study shows that the suppression of the stimulated immune response after CPB can be alleviated by iv administration of mannitol or hemofiltration. In the light of data showing that this depression of the immune response might affect the postoperative course of patients, these results could lead to an improvement of the management of patients undergoing cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* male patients
* aged 35-80
* elective CABG surgery

Exclusion Criteria:

* previous cardiac surgery
* ejection fraction < 40%
* valvular heart disease
* myocardial infarction during the last 3 months
* evidence of concomitant malignant or immunologic diseases
* antecedent medication with corticosteroids or methylxanthines
* hemoglobin < 12 g/dl
* body mass index > 30

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2003-10; Study Completion 2004-11

PRIMARY OUTCOMES:
LPS-stimulated cytokine release
LPS-stimulated CD14 exppression density

CONTACTS AND LOCATIONS:
Overall Officials: Hauke Rensing, MD PhD, Principal Investigator — University of Saarland
Locations (1):
- University of Saarland, Department of Anesthesiology, Intensive Care Medicine and Pain Therapy, Homburg/Saar, Saarland, Germany

REFERENCES:
- [Background] Wan S, LeClerc JL, Vincent JL. Inflammatory response to cardiopulmonary bypass: mechanisms involved and possible therapeutic strategies. Chest. 1997 Sep;112(3):676-92. doi: 10.1378/chest.112.3.676. PMID 9315800
- [Background] Grundmann U, Rensing H, Adams HA, Falk S, Wendler O, Ebinger N, Bauer M. Endotoxin desensitization of human mononuclear cells after cardiopulmonary bypass: role of humoral factors. Anesthesiology. 2000 Aug;93(2):359-69. doi: 10.1097/00000542-200008000-00013. PMID 10910482
- [Background] Wilhelm W, Grundmann U, Rensing H, Werth M, Langemeyer J, Stracke C, Dhingra D, Bauer M. Monocyte deactivation in severe human sepsis or following cardiopulmonary bypass. Shock. 2002 May;17(5):354-60. doi: 10.1097/00024382-200205000-00002. PMID 12022753
- [Background] Kleinschmidt S, Wanner GA, Bussmann D, Kremer JP, Ziegenfuss T, Menger MD, Bauer M. Proinflammatory cytokine gene expression in whole blood from patients undergoing coronary artery bypass surgery and its modulation by pentoxifylline. Shock. 1998 Jan;9(1):12-20. doi: 10.1097/00024382-199801000-00002. PMID 9466468
- [Background] Ziegenfuss T, Wanner GA, Grass C, Bauer I, Schuder G, Kleinschmidt S, Menger MD, Bauer M. Mixed agonistic-antagonistic cytokine response in whole blood from patients undergoing abdominal aortic aneurysm repair. Intensive Care Med. 1999 Mar;25(3):279-87. doi: 10.1007/s001340050836. PMID 10229162